CLINICAL TRIAL: NCT02557789
Title: A Study to Assess the Bioavailability and Pharmacokinetics of an Immediate Release Tablet Formulation of Lefamulin When Administered to Fed and Fasted Healthy Subjects in Comparison to an Intravenous Formulation and a Capsule Formulation
Brief Title: Bioavailability and Pharmacokinetics of Lefamulin When Administered to Fed and Fasted Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NAB-BC-3781-1107
Record Dates: First submitted 2015-07-27; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Absolute bioavailability; Pharmacokinetics
MeSH Terms: interventions — lefamulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment A (Experimental): Lefamulin as a 600 mg IR tablet in the fasted state
  Interventions: Drug: Lefamulin
- Treatment B (Experimental): Lefamulin as 600 mg API in capsule (three 200 mg capsules) in the fasted state
  Interventions: Drug: Lefamulin
- Treatment C (Experimental): Lefamulin as 150 mg i.v. in 250 mL citrate buffered saline infused over 1 h
  Interventions: Drug: Lefamulin
- Treatment D (Experimental): Lefamulin as a 600 mg IR tablet one hour after breakfast
  Interventions: Drug: Lefamulin

INTERVENTIONS:
Drug: Lefamulin — Lefamulin administered iv or orally in the fasted state and orally in the fed state
  Other Names: BC-3781

SUMMARY:
A Phase 1 study to assess the bioavailability and pharmacokinetics of a 600 mg immediate release tablet formulation of lefamulin when administered to fed and fasted healthy subjects in comparison to an intravenous formulation and a capsule formulation.

DETAILED DESCRIPTION:
This is a single center, single cohort, open label, randomized, four- period cross-over study with healthy subjects receiving a single dose of lefamulin at four study sessions at least 4 days apart. Lefamulin will be taken: 1) as 600 mg IR tablet orally in the fasted state; 2) as 600 mg API in capsule (3 x 200 mg capsules) orally in the fasted state; 3) as 150 mg i.v. infusion in 250 mL citrate buffered saline over 1 h; 4) as 600 mg IR tablet orally one hour after breakfast.

The order will be randomized. A total of 20 healthy subjects will be enrolled in the study. The same subjects will take part in all study sessions.

After each study session, the Safety Monitoring Team will review the safety and tolerance data before the commencement of the subsequent session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 18-55 years of age
* Good state of health (mentally and physically) as determined by the investigator
* Body mass index within the range 19 to 32 kg/m2 inclusive
* A signed and dated written informed consent form
* The subject is able to understand and willing to comply with protocol requirements and timetables, instructions and protocol-stated restrictions

Exclusion Criteria:

* Any acute or chronic illness or clinically relevant abnormality identified on the screening medical assessment, laboratory tests or ECG (12-lead or Holter), unless in the opinion of the investigator, in consultation with the Nabriva medical monitor, it will not interfere with the study procedures, affect the outcome of the study or compromise the safety of the subject
* A known history of chronic liver or biliary disease, history of Gilbert's syndrome or an elevated bilirubin level
* History of gastritis, gastrointestinal tract disorders or other clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of lefamulin
* Use of prescription or non-prescription drugs within 7 days or 10 times the elimination half-life (whichever is longer) prior to first dose of study medication
* Any intake of prescription or non-prescription drugs known to induce or inhibit drug-metabolizing enzymes or transport system enzymes within a period of less than 10 times the respective elimination half-life, or intake of grapefruit juice or grapefruit containing products within 7 days prior to first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The area under the concentration time curve (AUC) of an intravenous and oral formulation of lefamulin in the fasting state | 36 hours

SECONDARY OUTCOMES:
The area under the concentration time curve (AUC) of a tablet and capsule formulation of lefamulin in the fasting state | 36 hours
The area under the concentration time curve (AUC) of a 600 mg IR tablet of lefamulin in the fed state | 36 hours
Assessment of the safety and tolerability of lefamulin when administered, as single doses orally and i.v. to healthy subjects aged 18 to 55 years (adverse events, laboratory assessments, vital signs and electrocardiograms) | 36 hours
  Assessment of safety and tolerability by recording adverse events, laboratory assessments, vital signs and electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: William T Prince, MB, BChir, Study Chair — Nabriva Therapeutics AG
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom